M.03.RIC
INFORMATIVA E CONSENSO TRATTAMENTO DATI
SPERIMENTAZIONI CLINICHE
REV. 0 DEL 18/05/2021
PAGINA 1 DI 7

| DEMANGIT |
|----------|
| KEMAY-EH |

UOC Anestesia e Terapia Intensiva Donna Bambino Direttore UO: Dott. Giuseppe Sofi; Sperimentatore Principale: Dott.ssa Giovanna Chidini

# INFORMATIVA E MANIFESTAZIONE DEL CONSENSO AL TRATTAMENTO DEI DATI PERSONALI PER SPERIMENTAZIONI CLINICHE ai sensi dell'art. 13 del Regolamento n. 2016 / 679/ UE (GDPR) e della normativa privacy nazionale vigente

Versione n. 1 del 11/11/2021

"Reclutamento polmonare e ventilazione meccanica titolati con elettroimpedenziometria toracica nella sindrome da Distress Respiratorio Acuto in età pediatrica"

Gentile Signora/Signore,

questa informativa riguarda l'utilizzo dei dati personali, compresi i dati relativi alla salute e, se applicabile, di alcune categorie particolari di dati personali (es. dati genetici, dati rivelatori dell'orientamento e delle abitudini sessuali), per seguire obiettivi di ricerca in ambito scientifico.

## Finalità e natura del trattamento dei dati

La Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (da questo punto denominata Fondazione) è un Istituto di Ricovero e Cura a Carattere Scientifico le cui attività cliniche sono strumentali al perseguimento della ricerca scientifica.

Per partecipare ad uno studio clinico, è necessario che il soggetto aderente esprima, oltre al consenso per la partecipazione allo studio, anche il consenso al trattamento dei propri dati personali che potranno così essere utilizzati per perseguire obiettivi di ricerca utili per l'avanzamento delle conoscenze in campo scientifico.

I dati personali saranno trattati soltanto se sarà indispensabile in funzione della realizzazione degli obiettivi prefissati dallo Studio nonché, se applicabile, a fini di farmacovigilanza.

Il trattamento dei dati personali è indispensabile per lo svolgimento dello Studio; pertanto, un eventuale rifiuto di conferirli comporterà l'impossibilità di partecipare allo Studio.

# Promotore dello Studio

Il Promotore dello Studio è la Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico con sede legale a Milano, in via Francesco Sforza n. 28.

### Titolare del trattamento e Responsabile della protezione dei dati

Il Titolare del trattamento dei dati personali, comprese le categorie particolari di dati ai sensi dell'art. 9 GDPR, conferiti per l'esecuzione dello Studio che Le è stato presentato, è la Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, in qualità di Promotore dello Studio, con sede legale a Milano in via Francesco Sforza n. 28.

Il Responsabile della protezione dei dati (*DPO - Data Protection Officer*), nominato dalla Fondazione, in conformità all'art. 37 GDPR, potrà essere contattato scrivendo a dpo@policlinico.mi.it.





M.03.RIC INFORMATIVA E CONSENSO TRATTAMENTO DATI SPERIMENTAZIONI CLINICHE REV. 0 DEL 18/05/2021 PAGINA 2 DI 7

| REM | <b>A X 7</b> | CIT |
|-------|--------------|------|
| KEIVI | ΑV | -611 |

UOC Anestesia e Terapia Intensiva Donna Bambino Direttore UO: Dott. Giuseppe Sofi; Sperimentatore Principale: Dott.ssa Giovanna Chidini

## Soggetti ai quali potranno essere comunicati i dati personali

I dati personali raccolti dall'Unità Operativa che segue il paziente, saranno trasmessi al Promotore o, se del caso, alle società esterne incaricate di eseguire il monitoraggio e la verifica dello Studio. Pertanto, la partecipazione allo Studio implica che potranno venire a conoscenza dei dati, contenuti anche nella documentazione clinica originale, i seguenti soggetti (oltre a quelli indicati nel paragrafo precedente): il personale dell'Unità Operativa, il Comitato Etico e le autorità sanitarie italiane e straniere (es. AIFA, EMA, FDA). Questi ultimi esclusivamente ai fini del controllo delle procedure della sperimentazione e della correttezza ed esattezza dei dati raccolti, adottando, in ogni caso, tutte le cautele affinché venga garantita la necessaria riservatezza della identità del paziente e comunque nei limiti posti dalle norme applicabili, in particolare nello scrupoloso rispetto dei principi di correttezza, competenza, esattezza, pertinenza e completezza del trattamento.

I dati potranno essere altresì utilizzati per l'adesione da parte del Promotore a registri internazionali, in cui vengono conservati e condivisi dai ricercatori, in conformità al principio di scienza aperta (open science) e all'accesso libero ai dati della ricerca (open access), serie di dati (quali a titolo esemplificativo: sequenze di DNA, strutture proteiche, dati della ricerca preclinica e delle sperimentazioni cliniche, come pure dati epidemiologici). In tal caso i dati del paziente saranno condivisi in forma pseudonimizzata o anonimizzata, e saranno accessibili, tramite un apposito codice, solamente agli enti di ricerca che aderiscono ai suddetti registri internazionali.

# Tipologie di dati che potranno essere oggetto del trattamento

Per la conduzione dello Studio, potranno essere trattati, oltre ai dati personali del soggetto interessato (tra cui, a titolo esemplificativo, nome, età, etc..) anche categorie particolari di dati personali ai sensi dell'art. 9 GDPR, con particolare riferimento ai dati idonei a rivelare la salute del soggetto interessato nonché, se applicabile in base allo Studio, ai dati genetici, e ai dati idonei a rivelare l'orientamento e/o le abitudini sessuali.

#### Base giuridica del trattamento

I dati personali del soggetto aderente allo studio clinico saranno trattati sulla base di uno o più dei seguenti presupposti di liceità:

- Espressione del consenso esplicito dell'interessato (Art. 6.1, lett. a) e Art. 9.2, lett. a) GDPR;
- Salvaguardare gli interessi vitali dell'interessato e/o della collettività (Art. 6.1, lett. d) GDPR;
- Il trattamento è necessario per tutelare un interesse vitale dell'interessato o di un'altra persona fisica qualora l'interessato si trovi nell'incapacità fisica o giuridica di prestare il proprio consenso (Art. 9.2, lett. c) GDPR;
- Il trattamento è necessario per motivi di interesse pubblico nel settore della sanità pubblica, quali la protezione da gravi minacce per la salute a carattere transfrontaliero o la garanzia di parametri elevati di qualità e sicurezza dell'assistenza sanitaria e dei medicinali e dei dispositivi medici, sulla base del diritto dell'Unione o degli Stati membri che prevede misure appropriate e specifiche per tutelare i diritti e le libertà dell'interessato, in particolare il segreto professionale (Art. 9.2, lett. i) GDPR;
- Il trattamento è necessario ai fini di archiviazione nel pubblico interesse, di ricerca scientifica o storica o a fini statistici (Art. 9.2, lett. j) GDPR.





M.03.RIC DRMATIVA E CONS

Informativa e consenso trattamento dati sperimentazioni cliniche rev. 0 del 18/05/2021 pagina 3 di 7

| DΙ | ₹М. | AV. | PIT |
|-----|-------|----------------|-------|
| 1/1 | . ۲۷۱ | / <b>1</b> γ . | -1:11 |

UOC Anestesia e Terapia Intensiva Donna Bambino Direttore UO: Dott. Giuseppe Sofi; Sperimentatore Principale: Dott.ssa Giovanna Chidini

## Trasferimento dei dati a un Paese terzo o a un'organizzazione internazionale

Nel caso lo Studio preveda che i dati personali codificati vengano trasferiti e trattati in paesi al di fuori dell'Area Economica Europea (European Economic Area - EEA), la informiamo che in alcuni Paesi il livello di protezione dei dati potrebbe non essere ritenuto adeguato a quanto richiesto dalla Commissione Europea. Saranno, comunque, adottate tutte le misure di sicurezza appropriate per salvaguardare i diritti del soggetto in materia di riservatezza dei dati.

In particolare, il trattamento al di fuori del territorio dell'Area Economica Europea sarà ammesso solo se:

a) il Paese all'interno del quale avviene il trattamento ha un livello di protezione adeguato secondo gli standard previsti dalla Commissione Europea (ai sensi dell'art. 45 GDPR);

o se non vi è un'apposita dichiarazione della Commissione Europea sull'adeguatezza del Paese:

b) i dati personali saranno trattati nel rispetto delle appropriate garanzie di cui all'art. 46 GDPR, ad esempio tramite la sottoscrizione delle clausole standard approvate dalla Commissione Europea, ovvero sulla base di una delle deroghe previste dall'art. 49 GDPR, quali ad esempio, il consenso dell'interessato.

Maggiori informazioni sono disponibili presso il DPO, scrivendo agli indirizzi precedentemente indicati.

#### Conservazione dei dati personali

I dati personali raccolti nell'ambito di questo Studio verranno conservati presso l'Unità Operativa che ha in cura il paziente, presso il Promotore e presso le strutture coinvolte nello Studio, per il periodo di durata dello Studio come indicata nel Protocollo, ed eventuali proroghe che si rendessero eventualmente necessarie per la prosecuzione delle attività di ricerca. Tale termine potrà estendersi fino a un periodo massimo di 25 anni dopo la conclusione dello Studio, per ragioni connesse alla ricerca scientifica.

In particolare, il presente documento verrà archiviato conservato presso gli archivi della Fondazione, come da normativa vigente, mentre una copia integrale verrà consegnata al soggetto partecipante alla sperimentazione.

### Modalità del trattamento

Lo Sperimentatore e il suo staff che seguiranno il soggetto durante la sperimentazione tratteranno i dati personali, diversi da quelli identificativi (anagrafici), in modo da impedire di associarli in alcun modo al paziente, cioè trasmettendoli in forma pseudonimizzata. A tal fine, lo Sperimentatore assegnerà, all'inizio della sperimentazione, un codice con il quale identificherà il soggetto durante tutte le fasi della sperimentazione. I dati rilevanti per la sperimentazione, ad eccezione del nominativo del paziente, saranno registrati, elaborati e conservati unitamente a tale codice e a tutti i dati clinici inerenti lo stato di salute. Soltanto lo Sperimentatore e i soggetti autorizzati potranno collegare questo codice al nominativo del paziente.

I dati saranno trattati mediante strumenti informatici e non informatici ed archiviati in archivi cartacei e banche dati elettroniche e saranno diffusi solo in forma rigorosamente anonimizzata, ad esempio attraverso pubblicazioni scientifiche, statistiche e convegni scientifici.

Il Titolare del trattamento adotterà tutte le misure tecnico-organizzative per garantire il rispetto del principio di minimizzazione, come disposto dall'art. 80 GDPR.





M.03.RIC

Informativa e consenso trattamento dati sperimentazioni cliniche rev. 0 del 18/05/2021 pagina 4 di 7

| DEM | AXI DIT |
|--------|-----------|
| KEUVLA | 4 V-F.I I |

UOC Anestesia e Terapia Intensiva Donna Bambino Direttore UO: Dott. Giuseppe Sofi; Sperimentatore Principale: Dott.ssa Giovanna Chidini

#### Esercizio dei diritti

L'interessato ha i seguenti diritti:

- diritto di revoca del consenso in qualsiasi momento senza pregiudicare la liceità del trattamento basata sul consenso prestato prima della revoca, ex Art. 7, par. 3 GDPR;
- diritto di chiedere al Titolare del trattamento, ex Art. 15 GDPR, di poter accedere ai propri dati personali;
- diritto di chiedere al Titolare del trattamento, ex Art. 16 GDPR di poter rettificare i propri dati personali, ove quest'ultimo non contrasti con la normativa vigente sulla conservazione dei dati stessi e con la necessità di tutelare, in caso di contenzioso giudiziario, i professionisti sanitari che li hanno trattati;
- diritto di chiedere al Titolare del trattamento, ex Art. 17 GDPR, di poter cancellare i propri dati personali, ove quest'ultimo non contrasti con la normativa vigente sulla conservazione dei dati stessi e con la necessità di tutelare, in caso di contenzioso giudiziario, i professionisti sanitari che li hanno trattati;
- diritto di chiedere al Titolare del trattamento, ex Art. 18 GDPR, di poter limitare il trattamento dei propri dati personali;
- diritto di opporsi al trattamento, ex Art. 21 GDPR;
- diritto di chiedere al Titolare del trattamento, solamente nei casi previsti all'art. 20 del GDPR, che venga compiuta la trasmissione dei propri dati personali ad altro operatore sanitario in formato leggibile.

Infine, è riconosciuto il diritto di proporre reclamo all'Autorità di controllo incaricata della protezione dei dati, di cui all'art. 77 GDPR: Garante della privacy – email: garante@garanteprivacy.it.

Potrà esercitare i diritti sopra riportati:

- ✓ scrivendo al Titolare al seguente recapito: <u>privacy@policlinico.mi.it</u> oppure
- ✓ inviando una raccomandata a: Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, via Francesco Sforza n. 28, 20122 Milano all'attenzione del Titolare del trattamento.

Per esercitare il diritto di revoca è possibile compilare l'apposito spazio alla fine del presente documento e trasmetterlo attraverso le modalità sopra indicate.





M.03.RIC

INFORMATIVA E CONSENSO TRATTAMENTO DATI SPERIMENTAZIONI CLINICHE REV. 0 DEL 18/05/2021 PAGINA 5 DI 7

| REMAV-EIT |
|------------|
| IXEMIAY-EH |

UOC Anestesia e Terapia Intensiva Donna Bambino Direttore UO: Dott. Giuseppe Sofi; Sperimentatore Principale: Dott.ssa Giovanna Chidini

#### **DEFINIZIONI**

DATI PERSONALI: qualsiasi informazione riguardante una persona fisica identificata o identificabile («interessato»); si considera identificabile la persona fisica che può essere identificata, direttamente o indirettamente, con particolare riferimento a un identificativo come il nome, un numero di identificazione, dati relativi all'ubicazione, un identificativo online o a uno o più elementi caratteristici della sua identità fisica, fisiologica, genetica, psichica, economica, culturale o sociale.

DATI PARTICOLARI: dati personali che rivelano l'origine razziale o etnica, le opinioni politiche, le convinzioni religiose o filosofiche, o l'appartenenza sindacale; i dati genetici, i dati biometrici intesi a identificare in modo univoco una persona fisica, i dati relativi alla salute o alla vita sessuale o all'orientamento sessuale della persona.

DATI RELATIVI ALLA SALUTE: i dati personali attinenti alla salute fisica o mentale di una persona fisica, compresa la prestazione di servizi di assistenza sanitaria, che rivelano informazioni relative al suo stato di salute.

DATI GENETICI: i dati personali relativi alle caratteristiche genetiche ereditarie o acquisite di una persona fisica che forniscono informazioni univoche sulla fisiologia o sulla salute di detta persona fisica, e che risultano in particolare dall'analisi di un campione biologico della persona fisica in questione.

PSEUDONIMIZZAZIONE: il trattamento dei dati personali in modo tale che i dati personali non possano più essere attribuiti a un interessato specifico senza l'utilizzo di informazioni aggiuntive, a condizione che tali informazioni aggiuntive siano conservate separatamente e soggette a misure tecniche e organizzative intese a garantire che tali dati personali non siano attribuiti a una persona fisica identificata o identificabile.

TITOLARE DEL TRATTAMENTO: la persona fisica o giuridica, l'autorità pubblica, il servizio o altro organismo che, singolarmente o insieme ad altri, determina le finalità e i mezzi del trattamento di dati personali; quando le finalità e i mezzi di tale trattamento sono determinati dal diritto dell'Unione o degli Stati membri, il titolare del trattamento o i criteri specifici applicabili alla sua designazione possono essere stabiliti dal diritto dell'Unione o degli Stati membri.

RESPONSABILE DEL TRATTAMENTO: la persona fisica o giuridica, l'autorità pubblica, il servizio o altro organismo che tratta dati personali per conto del titolare del trattamento.

#### PRINCIPALI RIFERIMENTI GIURIDICI

- Regolamento Generale sulla Protezione dei Dati Personali UE 679/2016
- Codice in Materia di protezione dei dati Personali D.lgs. 101/2018
- Provvedimento 146/2019 dell'Autorità Garante della Privacy che individua prescrizioni relative al trattamento dei dati personali effettuati per scopi di ricerca scientifica
- Linea guida dell'European Data Protection Board 07/2020 che individuano prescrizioni relative al titolare e al responsabile del trattamento dei dati.

Il Titolare del trattamento (Promotore) Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico









M.03.RIC INFORMATIVA E CONSENSO TRATTAMENTO DATI SPERIMENTAZIONI CLINICHE REV. 0 DEL 18/05/2021

| REMAV-EIT |
|-----------|

PAGINA 6 DI 7

UOC Anestesia e Terapia Intensiva Donna Bambino

| Direttore UO: Dott. Giuseppe Sofi;<br>Sperimentatore Principale: Dott.ssa Giovani | na Chidini |
|---|---|
| <u>PRESA VISIONE DELL</u> | L'INFORMATIVA E MANIFESTAZIONE DEL CONSENSO |
| Cognome e nome del paziente | sesso M F |
| nato/a il/ / a | Recapito telefonico |
| Residente a | in via |
| L'informativa al trattamento dei dati persona | ali è stata presentata a: |
| Paziente | |
| Genitori (per i minori indicare i dati dei | due genitori) |
| Primo genitore: Cognome e Nome | nato il// |
| Secondo genitore: Cognome e Nome | nato il// |
| ☐ Tutore ☐ Amministratore of | <u> </u> |
| Cognome e Nome | nato il// |
| | n stampatello di chi esprime il consenso in caso di minore inserire i nomi di entrambi i genitori) |
| | DICHIARO |
| | evuto informazioni comprensibili ed esaurienti sul trattamento dei dati proposto. Valutate le informazioni ricevute: |
| ☐ ACCONSENTO | ☐ NON ACCONSENTO |
| al trattamento dei dati personali, compres<br>nei limiti e con le modalità indicate nell'in | si i dati relativi alla salute, e al loro trasferimento per le finalità dello Studio,<br>formativa. |
| ACCONSENTO | ☐ NON ACCONSENTO |
| alla condivisione dei dati personali come s<br>limiti e nelle modalità indicate nell'inform | sopra identificati, per l'adesione del Promotore a registri internazionali, nei ativa. |
| Data / / | Firma del paziente/genitori/tutore/amministratore di sostegno |

ISTITUTO DI RICOVERO E CURA A CARATTERE SCIENTIFICO DI NATURA PUBBLICA Via Francesco Sforza, 28 - 20122 Milano Tel. 02 5503.1 - www.policlinico.mi.it - CF e P.I. 04724150968









#### M.03.RIC

INFORMATIVA E CONSENSO TRATTAMENTO DATI
SPERIMENTAZIONI CLINICHE
REV. 0 DEL 18/05/2021
PAGINA 7 DI 7

| REMAV-EIT |
|-----------|
|-----------|

UOC Anestesia e Terapia Intensiva Donna Bambino Direttore UO: Dott. Giuseppe Sofi; Sperimentatore Principale: Dott.ssa Giovanna Chidini

| REVOCA DEL CONSENSO | |
|---|---|
| lo sottoscritto/a (cognome e nome) | nato/a il |
| revoco il consenso precedentemente espresso. Sono consapevole che l'esercizio del mio diritto di revoca comport l'immediata cancellazione dei dati forniti in precedenza e la conseguente interruzione della partecipazione allo studio clinico, non pregiudicando la liceità dei trattamenti eseguiti fino a questo momento. | |
| Data/ Firms | a del paziente/genitori/tutore/amministratore di sostegno |





